CLINICAL TRIAL: NCT00702598
Title: The WORKER Study: A Randomized Controlled Trial of Escitalopram and Telephone-based Cognitive Behaviour Therapy in Working Patients With Major Depressive Disorder
Brief Title: The WORKER Study: Escitalopram and Telephone-based Cognitive Behaviour Therapy (CBT) for Depressed Working People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H07-03029
Record Dates: First submitted 2008-06-18; First posted 2008-06-20 (Estimated); Last update posted 2012-05-09 (Estimated); Status verified 2012-05

CONDITIONS: Major Depressive Disorder (MDD)
Keywords: Depression; occupational function; rating scales; RCT; cognitive behaviour therapy; CBT; escitalopram; antidepressants
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Telephone-based Cognitive Behaviour Therapy
  Interventions: Behavioral: Telephone-based Cognitive Behaviour Therapy (CBT)
- 2 (Placebo Comparator): Telephone reminder calls
  Interventions: Behavioral: Telephone reminder calls

INTERVENTIONS:
Behavioral: Telephone-based Cognitive Behaviour Therapy (CBT) — Telephone-based CBT: Eight sessions of telephone-based CBT (Tel-CBT) will be delivered over 8-10 weeks, based on a published manual (Simon et al, 2004). Tel-CBT has been modified to be briefer than traditional CBT (30-40 minutes instead of 60 minutes per session) and will be offered at convenient times (including evening sessions). The initial Tel-CBT session will occur within 2 weeks of randomization, with subsequent sessions occurring every 1-2 weeks depending on scheduling and patient preference. The initial session focuses on motivation enhancement exercises, subsequent sessions emphasize identifying, challenging and distancing from negative thoughts, and the final session focuses on a personal care plan and self-management skills.
  Arms: 1
Behavioral: Telephone reminder calls — Telephone reminder calls: Weekly telephone calls for 8 weeks to inquire on progress and remind patients to take their medications properly
  Arms: 2

SUMMARY:
This study will investigate the additional benefits of telephone-based cognitive behavioral therapy (Tel-CBT) as added treatment to an antidepressant (escitalopram) in working people with major depressive disorder (MDD) versus treatment with escitalopram alone. Outcomes will include depression symptom rating scales and measures of work absence and productivity. The hypothesis is that Tel-CBT and escitalopram will result in better outcomes than escitalopram alone in working patients with MDD.

DETAILED DESCRIPTION:
Rationale CBT is recognized as an effective psychological treatment for MDD. However, there are still considerable barriers to access CBT. Newer methods of delivering CBT, such as over the telephone (Tel-CBT), allow for greater access and convenience, at potentially lower cost. This is especially relevant for working people because the service can be delivered during evenings and weekends, so they do not need to leave work to attend clinic appointments. Ease of access is also important for rural settings where distance to health facilities can be a barrier to care. The ease of delivery of Tel-CBT, both in setup and maintenance costs, may also make it an important component of enhanced support for primary care. Preliminary studies have shown that addition of Tel-CBT leads to better outcomes than usual care alone (Simon et al, 2004; Wang et al, 2007).

This study will investigate the added value of Tel-CBT as adjunctive treatment to an antidepressant (escitalopram) in working people with MDD versus treatment with escitalopram alone, focusing on work-related outcomes. Escitalopram offers advantages as a first-choice treatment for depressed working people, given its superior efficacy compared to other antidepressants, excellent tolerability and simplicity of use for family physicians. Observational studies have shown significant reductions in sick leave when depressed patients are treated with escitalopram (Winkler et al, 2007). Outcome will be rigorously evaluated by assessing absenteeism and work productivity, response and remission rates, and quality of life, after acute (3 month) treatment and longer-term (6 month) follow-up.

Research Method This is a 6-month, multi-centre, single-blind (rater), randomized, parallel-design study to assess the efficacy of escitalopram and Tel-CBT in the treatment of working subjects with MDD, compared to treatment with escitalopram alone. A total of 150 depressed patients meeting entry criteria will be enrolled over a 1 year period.

Eligible patients will be treated with escitalopram 10-20 mg/d for the entire treatment period (6 months). Patients will be randomized to addition of telephone-based CBT with 8 sessions conducted over a 3 month period, or to a (placebo) control condition of reminder telephone calls. Outcomes (HAM-D, MADRS) will be primarily assessed over the telephone by raters blind to treatment assignment. Other outcome measures will be assessed by patient-rated questionnaires administered over the internet using a secure web site, and by ratings from the treating physician (CGI and adverse events).

Statistical Analysis All randomized subjects who have at least one follow-up visit will be included in the analysis based on intent-to-treat. Ineligible subjects who are inappropriately randomized will be excluded from the analysis. Missing data will be imputed using last observation carried forward (LOCF). For the analyses the treatment variables will remain coded and the analysts and investigators will remain blinded to variable identity during analysis and interpretation.

The pre-specified primary efficacy endpoint is the adjusted mean change from baseline to endpoint (12 weeks) in the HAM-D score using LOCF. All comparisons will be analyzed using ANCOVA adjusting for baseline value and centre. The secondary outcomes will also be analyzed using a similar analysis, when appropriate. Post hoc analyses will also examine observed case data. Categorical data (such as proportions of the sample with adverse events) will be analyzed using chi-square tests or Fisher's test where cell sizes warrant.

ELIGIBILITY:
Inclusion Criteria:

* Male and female outpatients aged 18-65 years.
* Patients will meet DSM-IV criteria for major depressive disorder as determined by the mood disorders section of the Mini International Neuropsychiatric Interview (MINI, Sheehan et al, 1998).
* Currently employed (or off work for 2 weeks or less, and expecting to return to work at the start of study).
* A score of 18 or greater on the self-rated version of the MADRS, indicating at least moderately severe depression.
* Competency to give informed consent.

Exclusion Criteria:

* Patients on short-term (except for circumstances under Inclusion Criteria) or long-term disability.
* Pregnant women, lactating women and sexually active women of childbearing potential who are not using medically accepted means of contraception.
* Serious suicidal risks as judged by the study doctor.
* The following DSM-IV diagnoses (to ensure a homogenous diagnostic group): Organic mental disorders; Substance abuse/dependence, including alcohol, active within the last year; Schizophrenia, Paranoid or Delusional Disorders; Other Psychotic disorders; Panic disorder; Generalized Anxiety Disorder; Obsessive-Compulsive Disorder, or Post Traumatic Stress Disorder, if a primary diagnosis; Bipolar Disorder;Bulimia Nervosa; Anorexia Nervosa.
* Serious illness including cardiac, hepatic, renal, respiratory, endocrinologic, neurologic and hematologic disease that is not stabilized.
* Regular or current use of other psychotropic drugs.
* Use of monoamine oxidase inhibitors within 14 days of Visit 1, fluoxetine within 5 weeks of Visit 1, and other antidepressants within 7 days of Visit 1 (to ensure adequate drug washouts prior to starting escitalopram).
* Previous use of escitalopram.
* Treatment resistance in the current episode, as defined by failure (lack of clinically significant response) of two or more antidepressants given at therapeutic doses for at least 6 weeks.
* Patients who start formal psychotherapy (e.g. cognitive-behavioural or interpersonal psychotherapy) within 3 months of Visit 1, or who plan to initiate such psychotherapy during this study.
* Patients involved in any other form of treatment for depression.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2008-06; Primary Completion 2011-04 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Change in adjusted HAM-D and MADRS scores at 3 month followup | 6 months

SECONDARY OUTCOMES:
At 3 and 6 month followup: clinical response and remission rates, absenteeism and work productivity, adverse events, quality of life, and cost-effectiveness. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Raymond W. Lam, MD, FRCPC, Principal Investigator — University of British Columbia; Sagar V. Parikh, Study Director — University of British Columbia; Erin E. Michalak, Study Director — University of British Columbia; Kevin Solomons, Study Director — University of British Columbia; Sidney H. Kennedy, Ph.D, Study Director — University of British Columbia; Edwin M. Tam, Study Director — University of British Columbia
Locations (1):
- UBC Hospital Mood Disorders Centre, Vancouver, British Columbia, Canada

REFERENCES:
- [Background] Simon GE, Ludman EJ, Tutty S, Operskalski B, Von Korff M. Telephone psychotherapy and telephone care management for primary care patients starting antidepressant treatment: a randomized controlled trial. JAMA. 2004 Aug 25;292(8):935-42. doi: 10.1001/jama.292.8.935. PMID 15328325
- [Background] Wang PS, Simon GE, Avorn J, Azocar F, Ludman EJ, McCulloch J, Petukhova MZ, Kessler RC. Telephone screening, outreach, and care management for depressed workers and impact on clinical and work productivity outcomes: a randomized controlled trial. JAMA. 2007 Sep 26;298(12):1401-11. doi: 10.1001/jama.298.12.1401. PMID 17895456
- [Background] Winkler D, Pjrek E, Moser U, Kasper S. Escitalopram in a working population: results from an observational study of 2378 outpatients in Austria. Hum Psychopharmacol. 2007 Jun;22(4):245-51. doi: 10.1002/hup.839. PMID 17443491
- [Derived] Lam RW, Parikh SV, Ramasubbu R, Michalak EE, Tam EM, Axler A, Yatham LN, Kennedy SH, Manjunath CV. Effects of combined pharmacotherapy and psychotherapy for improving work functioning in major depressive disorder. Br J Psychiatry. 2013 Nov;203(5):358-65. doi: 10.1192/bjp.bp.112.125237. Epub 2013 Sep 12. PMID 24029535